CLINICAL TRIAL: NCT01200719
Title: Transcranial Alternating Current Stimulation (tACS) Enhances Neurological Function Recovery Among Post-stroke Patients
Brief Title: Transcranial Alternating Current Stimulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Yongshan Hu, Head of Rehabilitation Center, Huashan Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-102
Record Dates: First submitted 2010-09-10; First posted 2010-09-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2006-10

CONDITIONS: Stroke
Keywords: brain electrical stimulation; sub-acute post-stroke; rehabilitation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tACS group (Experimental)
  Interventions: Device: transcranial alternating current stimulation (tACS)
- Control group (No Intervention): Patients in the control group followed exactly the same protocol but without receiving the transcranial alternating current stimulation .

INTERVENTIONS:
Device: transcranial alternating current stimulation (tACS) — Patients in the tACS group received a total of 15 sessions of brain stimulation. The sessions were conducted on weekdays (from Monday to Friday) for three consecutive weeks. Each session lasted 30 minutes. The alternating current stimulations were generated by a CVFT-MG201 machine. Stimulations were delivered by two U-shaped electrodes (approximately 7 cm2) fixed on the patient's left and right mastoid regions (anode or cathode varied depending on polarity of the alternating current). The frequencies (supra-slow waves: < 1 Hz; theta to gamma), levels of intensities (0 to 3mA), and density function (follows a bell-shaped curve; mean intensity ~ 2.1mA) of the current were delivered according to the manufacturer's pre-set random protocol.
  Other Names: CVFT-MG201(China Patent No. ZL98121951.9)
  Arms: tACS group

SUMMARY:
To investigate the efficacy of using transcranial alternating current stimulation (tACS) to enhance the regaining of neurological function among post-stroke patients.

DETAILED DESCRIPTION:
Sixty post-stroke patients were randomly assigned to receive 15 sessions of the usual rehabilitation programme with or without tACS. The NIH Stroke Scale (NIHSS) and the mean blood flow velocity (MFV) and Gosling pulsatility index (PI) captured for the middle, anterior, and posterior cerebral artery were the outcome measures.

Fifteen 30-minute sessions of tACS appear to be effective for enhancing post-stroke patients' neurological function. The haemodynamic measures taken indicated that the regaining of function among the patients was largely attributed to a lowering of the vascular autoregulatory activity together with an increase in blood flow velocity at the middle cerebral artery. Future studies should explore the underlying mechanisms mediating the positive effects brought about by tACS in post-stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as first onset intracerebral haemorrhage or infarction (according to ICD-10 I61.0-I61.6 or I63.3-I63.6, with or without I69, i.e.: sequelae of cerebrovascular disease)
* between 15 and 60 days after the onset
* right handedness
* no previous neurological or psychiatric disorders
* positive transtemporal windows for bilateral middle, anterior, and posterior cerebral arteries insonation (according to the standards set by the Transcranial Doppler Ultrasonographic Device (TCD))
* NIH Stroke Scale (NIHSS) scores between 14 and 24
* not receiving rehabilitation before admission

Exclusion Criteria:

* medical comorbidity preventing the patient undergoing the intervention
* preceding epileptic fits
* having metallic implants in the brain or a pacemaker
* history of surgery to the brain

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2006-11; Primary Completion 2007-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
NIH Stroke Scale (NIHSS) score | 3 weeks

SECONDARY OUTCOMES:
the mean blood flow velocity (MFV) | 30 minutes
  captured for the middle, anterior, and posterior cerebral artery by transcranial Doppler
Gosling pulsatility index (PI) | 30 minutes
  captured for the middle, anterior, and posterior cerebral artery by transcranial Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Yongshan Hu, MD, Principal Investigator — Rehabilitation Center, Huashan Hospital of Fudan University, Shanghai, China; Chetwyn Chan, PhD, Study Director — Department of Rehabilitation Science, the Hong Kong Polytechnic University
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China